CLINICAL TRIAL: NCT06246383
Title: Effectiveness of Standardised Ido-BR1 Cucumber Extract (Q-ActinTM) on Mild to Moderate Joint Pain: A Randomized Double-blind Placebo-Controlled Study
Brief Title: Effectiveness of Cucumber Extract on Joint Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jacksonville University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: JacksonvilleU
Record Dates: First submitted 2024-01-22; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Joint Pain
MeSH Terms: conditions — Arthralgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QActin (Active Comparator): Cucumber extract
  Interventions: Dietary Supplement: Q Actin
- placebo (Placebo Comparator): Placebo capsule
  Interventions: Dietary Supplement: Q Actin

INTERVENTIONS:
Dietary Supplement: Q Actin — cucumber extract

SUMMARY:
Joint pain is reported by about 1/3 of U.S. adults, and increases with age reaching 50% prevalence among the elderly [1]. Joint pain is associated with substantial activity limitation, work disability, sleep disturbance, negative mood (e.g., depression, anxiety, stress), and reduced quality of life (2, 3).

Conventional treatment of joint pain with non-steroidal anti-inflammatory drugs (NSAIDs) and other analgesics is associated with gastrointestinal and cardiovascular side effects, and other adverse health effects [4]. Use of alternative supplements is reported by about 50% of people with knee osteoarthritis, and well-designed human trials are needed to identify effective analgesic alternatives [5]. The most widely used and studied joint pain supplements include those related to chondroprotection such as glucosamine, chondroitin, collagen hydrolysates, and hyaluronic acid [6-9]. Further research is needed examining the effects of other herbal supplementation on joint pain and overall health.

Preliminary research reveals Q-ActinTM supplementation may be an effective intervention to reduce OA-related pain compared with standard treatments. Q-ActinTM is a cucumber extract with the anti-inflammatory iminosugar idoBR1 standardised to over 1%.

Study Purpose To conduct a 8 week randomized double-blind placebo-controlled trial to examine the effectiveness of daily use of Q-ActinTM supplementation compared to placebo on joint pain, stiffness, function, mood, sleep, daytime activity, and health-related quality of life in adults with a history (>3 months) of mild to moderate joint pain.

DETAILED DESCRIPTION:
To conduct a 8 week randomized double-blind placebo-controlled trial to examine the effectiveness of daily use of Q-ActinTM supplementation compared to placebo on joint pain, stiffness, function, mood, sleep, daytime activity, and health-related quality of life in adults with a history (>3 months) of mild to moderate joint pain.

Assessments will be completed at Day 0 (Baseline), Week 2, Week 4, and Week 8. The primary outcome will be on joint pain, stiffness, and function (as assessed by the WOMAC). Secondary outcomes will be sleep quality, physical activity, daytime fatigue, mood, anxiety, perceived stress, pain severity, tolerance and limitations, and health-related quality of life.

Adults (N = 80) will be randomized to one of the following conditions:

* Q-ActinTM (n = 40)
* Placebo control (n = 40)

ELIGIBILITY:
Inclusion Criteria:

Inclusion and Exclusion Criteria: Participants (N = 80) will meet the inclusion criteria if they: are healthy adults (age range between 35 to 70 years), chose to sign Sterling IRB approved consent forms, and willing to forego use of all supplement products with claims regarding joint health during the study period. Our goal is to have 80 participants complete the intervention. To control for potential dropout we will recruit 90 participants for this trial.

Other inclusion and exclusion criteria for this study included:

1. Self-reported history (>3 months) of joint pain in the knees, hip, ankles, shoulders, or hands. Minimum symptom severity was ensured by using a WOMAC pain index score of at least 2 points.
2. No history of regular NSAID use (e.g., ibuprofen, aspirin) during the previous two weeks, and willingness to avoid NSAIDs use during the 8-week study.
3. Not on other medications (e.g., analgesic gels, arthritis medications, other anti-inflammatory drugs) or supplements (in particular, glucosamine and chondroitin) for joint pain for the previous two weeks, and willing to avoid use of these during the 8-week study.
4. No serious medical problems (current cancer case, severe rheumatoid arthritis, recent heart attack, recent stroke, congestive heart failure, ulcers, kidney disease, or other disease that would interfere with study participation).
5. No psychiatric disorder or other condition that might interfere with self-assessment ability.
6. Willingness to follow all study procedures including randomization to one of two groups, and to stay weight stable during the study.
7. Able to walk for at least 6 min at a moderate-to brisk pace.
8. No history of allergic reactions to shellfish products or products containing aspirin.
9. Pregnant or trying to conceive. Note: Paracetamol (i.e., acetaminophen as found in Tylenol) will be allowed as a rescue medicine for pain during the study as needed, with usage recorded.

   -

   Exclusion Criteria:

   -

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Joint pain | 8 weeks
  WOMAC

SECONDARY OUTCOMES:
mood, sleep, daytime activity, pain perceptions, daytime fatigue, anxiety, perceived stress, pain perceptions, health-related quality of life. | 8 weeks
  POMS, PSQI, Oura Ring, Daytime Fatigue Scale, Perceived Stress Scale, Trait Anxiety Scale, Pain Severity Scale, Health-related Quality of Life Scale

IPD SHARING:
Plan to Share IPD: Yes
Only group data will be shared
Supporting Information: Study Protocol, SAP
Time Frame: Summer 2024
Access Criteria: written request

REFERENCES:
- [Derived] Hausenblas HA, Hooper D, Hooper S. Effectiveness of Cucumis sativus L. Supplementation on Mood, Anxiety, and Sleep Quality: A Randomized Double-Blind Placebo-Controlled Study. Health Sci Rep. 2025 Jul 9;8(7):e70979. doi: 10.1002/hsr2.70979. eCollection 2025 Jul. PMID 40636535